CLINICAL TRIAL: NCT02645396
Title: A Cohort Study of Congenital Cytomegalovirus Infection Among Pregnant Women and Their Neonates in China
Brief Title: A Cohort Study of Congenital Cytomegalovirus Infection Among Pregnant Women and Their Newborns in China
Status: Completed | Type: Observational
Sponsor: Jun Zhang (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor-Investigator, Jun Zhang, Vice dean of School of Public Health,Xiamen University, Xiamen University
Organization: Xiamen University (Other)
Other Study IDs: CMV-EPI-001
Record Dates: First submitted 2015-07-31; First posted 2016-01-01 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Congenital Cytomegalovirus Infection; Cytomegalovirus Infection Reactivation
Keywords: Cytomegalovirus
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood/urine samples of the pregnant women; saliva /urine samples of the newborns
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the risk of congenital cytomegalovirus (cCMV) infection in newborns born to seropositive women.

DETAILED DESCRIPTION:
This study will be conducted at several Maternal and Child Health Hospitals (MCHHs) in China and the research activities will be integrated with routine medical services during pregnancy at the study sites.The investigators will build a perspective cohort study enrolling ~8000 pregnant women elder than 18 and following up their newborns at specific MCHHs.As a first step, The investigators will work with these hospitals to recruit the subjects. After being informed, the participants' remaining blood and urine samples (after their medical examinations) at their early, medium and late stages of pregnancy will be collected , and their newborns' urine and saliva samples will be collected after delivery. The aim of this study is to enroll 5000 series mother-newborns.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 and older
* Pregnancy confirmed by ultrasound
* Come to MCHHs for "Pregnancy Registry" within 24 weeks of pregnancy

Exclusion Criteria:

* Not capable of complying with study procedures, or having a psychosis, two-stage affective psychosis, or have a tendency to suicide
* Having any autoimmune diseases (include systemic lupus erythematosus, rheumatoid arthritis), immunodeficiency (e.g. AIDS), chronic disease history such as cancers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll ~8000 pregnant women aged 18 years and above at MCHHs. Pregnant women who meet the inclusion/exclusion criteria will be enrolled. All inclusion and exclusion criteria will be reviewed by investigators or qualified designees to ensure that each subject is qualified for the study. In general, those whose newborns (including early birth, any congenital anomaly) are successfully followed up remain in the study population. However, those with adverse pregnancy outcomes captured in the MCHHs, such as abortion and still birth, etc., will also be the investigators' subjects even though we cannot have newborns' urine/saliva samples.
Sampling Method: Probability Sample
Enrollment: 8855 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Incidence of cCMV infection in newborns born to CMV seropositive pregnant women. | up to 45 months

SECONDARY OUTCOMES:
Incidence of cCMV infection in newborns to pregnant women with different maternal PP150-IgG titers in the early pregnancy. | up to 45 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Professor, Principal Investigator — Xiamen University
Locations (2):
- China (2):
  - Maternity and Child care of Huli District, Xiamen, Fujian
  - Maternity and Child care of Xinmi City, Zhengzhou, Henan

REFERENCES:
- [Derived] Huang Y, Li T, Yu H, Tang J, Song Q, Guo X, Wang H, Li C, Wang J, Liang C, Yao X, Qiu L, Zhuang C, Bi Z, Su Y, Wu T, Ge S, Zhang J. Maternal CMV seroprevalence rate in early gestation and congenital cytomegalovirus infection in a Chinese population. Emerg Microbes Infect. 2021 Dec;10(1):1824-1831. doi: 10.1080/22221751.2021.1969290. PMID 34392819